CLINICAL TRIAL: NCT01217827
Title: Implantable Cardioverter-Defibrillator (ICD) Utilization in a Potentially Eligible VA Population
Brief Title: Implantable Cardioverter-Defibrillator Use in the VA System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Medtronic (Industry); VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul A. Heidenreich, Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SU-08102010-6708; IRB 15312
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Results first posted 2016-12-07 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Cardiomyopathies
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Clinical Reminder (Experimental): Reminder of potential candidacy for an implantable cardioverter defibrillator. The reminder is placed in the medical record with copy to the primary provider and any cardiologist managing the patient.
  Interventions: Behavioral: Clinical Reminder
- Control (No Intervention): This group does not receive an intervention.

INTERVENTIONS:
Behavioral: Clinical Reminder
  Arms: Clinical Reminder

SUMMARY:
Despite being a proven life-saving intervention in appropriately selected individuals, multiple studies continue to demonstrate low implantation of defibrillators in potential candidates. Based upon prior research, a major barrier to low utilization is low referral of potential candidates by healthcare providers. In this study, via brief clinical reminder placed in the electronic medical record, we ask healthcare providers who have not referred potential candidates for defibrillator the reasons for this decision and provide them with the tools for referral if appropriate.

ELIGIBILITY:
Inclusion Criteria:Meeting published criteria for receipt of an implantable cardioverter defibrillator Exclusion Criteria:provider is not affiliated with the VA health care system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Heidenreich, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, California
  - Stanford University School of Medicine, Stanford, California

REFERENCES:
- [Derived] Gupta A, Gholami P, Turakhia MP, Friday K, Heidenreich PA. Clinical reminders to providers of patients with reduced left ventricular ejection fraction increase defibrillator referral: a randomized trial. Circ Heart Fail. 2014 Jan;7(1):140-5. doi: 10.1161/CIRCHEARTFAILURE.113.000753. Epub 2013 Dec 6. PMID 24319096

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinical Reminder: Reminder of potential candidacy for an implantable cardioverter defibrillator. The reminder is placed in the medical record with copy to the primary provider and any cardiologist managing the patient.
  Clinical Reminder
Period: Overall Study
Arm/Group | Clinical Reminder | Control
Started | 46 | 43
Completed | 46 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinical Reminder | Control | Total
Number analyzed (Participants) | 46 | 43 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (8) | 64 (8) | 65 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 43 | 43 | 86
Region of Enrollment [Number; unit: participants]
  United States | 46 | 43 | 89

OUTCOME MEASURES:

1. Primary Outcome: Referral for Implantable Cardioverter Defibrillator
Description: Referral of the patient to electrophysiology clinic for evaluation for cardioverter defibrillator implantation.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Clinical Reminder | Control
Number analyzed (Participants) | 46 | 43
participants | 11 | 1

ADVERSE EVENTS:
Arm/Group | Clinical Reminder | Control
Serious Adverse Events (participants affected / at risk) | 1/46 | 4/43
Other Adverse Events (participants affected / at risk) | 0/46 | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinical Reminder (N=46) | Control (N=43)
Death (Cardiac disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes